CLINICAL TRIAL: NCT00622804
Title: Phase III Study on Comparison for Bile Reflux and Gastric Stasis in Patients With Gastric Cancer After Distal Gastrectomy
Brief Title: Comparison Study for Bile Reflux and Gastric Stasis in Patients After Distal Gastrectomy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: It was very difficult to enroll patients in this study.
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Wook Kim, Department of Surgery, Holy Family Hospital, College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCHC06OT049
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Stomach Cancer; Gastrectomy
Keywords: Stomach cancer; Gastrectomy; Postgastrectomy syndrome
MeSH Terms: conditions — Stomach Neoplasms; Postgastrectomy Syndromes | interventions — Gastroenterostomy; Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Billroth-II (B-II)reconstruction
  Interventions: Procedure: Billroth-II (B-II)
- 2 (Other): Roux en Y gastrojejunostomy (RY-GJ)
  Interventions: Procedure: Roux en Y gastrojejunostomy (RY-GJ)
- 3 (Other): uncut Roux en Y gastrojejunostomy (uncut RY-GJ)
  Interventions: Procedure: uncut Roux en Y gastrojejunostomy

INTERVENTIONS:
Procedure: Billroth-II (B-II) — After conventional distal gastrectomy with lymphadenectomy, jejunum of a distal segment from 10 to 20cm from Treitz is used for reconstruction. Jejunal segment is transposed in a way of ante-colon, and then gastrojejunostomy is performed using 60mm linear cutting stapler or hand-sawing technique with absorbable suture. After anastomosis, reinforcement suture is done.
  Other Names: B-II
  Arms: 1
Procedure: Roux en Y gastrojejunostomy (RY-GJ) — After conventional distal gastrectomy with lymphadenectomy, jejunum is transected in the segment from 10 to 20 cm, and then distal end is transposed in a way of retro-colon to perform anastomosis using 60mm linear cutting stapler or hand-sawing technique with absorbable suture. After anastomosis, reinforcement suture is done. The resected proximal jejunum and the portion of jejunum distal 45 cm from gastrojejunostomy are anastomosed using 60mm linear cutting stapler or hand-sawing technique with absorbable suture followed by reinforcement suture.
  Other Names: RY-GJ
  Arms: 2
Procedure: uncut Roux en Y gastrojejunostomy — After conventional distal gastrectomy with lymphadenectomy, jejunum of distal segment 45 cm from Treitz ligament is used for reconstruction. Jejunal segment is transposed in a way of ante-colon, and then gastrojejunostomy is performed using 60mm linear cutting stapler or hand-sawing technique with absorbable suture followed by reinforcement suture. After anastomosis, afferent loop distal 5cm is obstructed using non-cutting stapler or hand sawing suture. And then, distal jejunum 10 cm from obstructive portion and efferent jejunal loop distal 45 cm from gastrojejunostomy are anastomosed in a manner of side to side followed by reinforcement suture.
  Other Names: uncut RY-GJ
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the degree of bile reflux and gastric stasis according the reconstruction methods after distal subtotal gastrectomy for gastric cancer, and to find out the proper method. We collect ninety patients who undergo distal gastrectomy for gastric cancers for this study from 5 institutions and randomly divide into 3 groups according to reconstruction methods: 1) Billroth-II (B-II), 2) Roux en Y gastrojejunostomy (RY-GJ) and 3) uncut Roux en Y gastrojejunostomy (uncut RY-GJ).

DETAILED DESCRIPTION:
Patients who have undergone gastrectomy for gastric cancer might be developed various symptoms by gastric stasis and bile reflux, it so called "post-gastrectomy syndrome", because of the diminishment of stomach capacity, the decrease of expulsive ability and the change of food passage. Until now, that had been accepted as the inevitable results after gastric resection. However, the survival rate has recently been increased owing to the increased proportion of early gastric cancer. And thus, to improve the quality of life of patients, many researchers have been actually studying for the reconstruction methods which are able to minimize the symptom by gastrectomy, but it is dissatisfied until now. Thus, the purpose of this study is to evaluate the degree of bile reflux and gastric stasis according the reconstruction methods after distal subtotal gastrectomy for gastric cancer, and to find out the proper method.

We collect ninety patients who undergo distal gastrectomy for gastric cancers for this study from 5 institutions and randomly divide into 3 groups according to reconstruction methods: 1) Billroth-II (B-II), 2) Roux en Y gastrojejunostomy (RY-GJ) and 3) uncut Roux en Y gastrojejunostomy (uncut RY-GJ). We evaluate the postoperative morbidity rate and then the degree of bile reflux, gastric emptying time and quality of life through long term follow-up using the gastrofiberscope, survey and so on.

From this study, we would suggest the standard reconstruction procedure after distal gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent distal gastrectomy for adenocarcinoma of stomach with following criteria:

  1. have cancer located in middle or distal portions
  2. preoperative staged as cT1N0M0 or cT2N0M0 by computed tomography and gastrofiberscope (Endoscopic ultrasound, optionally)
  3. have The American Society of Anaesthesiologists (ASA) score of three and less

Exclusion Criteria:

* Patients following criteria:

  1. have simultaneously other cancer
  2. underwent cancer therapy (radiologic or immunologic or chemotherapeutic method) at past time
  3. have systemic inflammatory disease
  4. have upper gastrointestinal surgery
  5. have the gastric cancer with obstruction
  6. get pregnancy
  7. are treating diabetics with Insulin
  8. are participating or participated within 1 month in other clinical trials
  9. have BMI less than 25
  10. are expected to perform laparoscopy assisted gastrectomy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Bile reflux by Dual scintigraphy | six month and one year after operation

SECONDARY OUTCOMES:
Gastric emptying time by Dual scintigraphy | six month and one year after operation
Residual food, gastritis, bile reflux and reflux esophagitis by Gastrofiberscope findings | six month and one year after operation
Quality of life by EORTC QLQ30, STO22 | one year after operation
Morbidity and Mortality | In hosipital

CONTACTS AND LOCATIONS:
Overall Officials: Wook Kim, MD, PhD, Principal Investigator — Department of Surgery, Holy Family Hospital, The Catholic University of Korea
Locations (5):
- South Korea (5):
  - Department of Surgery, Holy Family Hospital, The Catholic University of Korea, Bucheon-si
  - Department of Surgery, Our Lady of Mercy Hospital, The Catholic University of Korea, Incheon
  - Department of Surgery, Kangnam St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Department of Surgery, St Mary's Hospital, The Catholic University of Korea, Seoul
  - Department of Surgery, St. Vincent's Hopital, The Catholic University of Korea, Suwon

REFERENCES:
- [Background] Ogoshi K, Okamoto Y, Nabeshima K, Morita M, Nakamura K, Iwata K, Soeda J, Kondoh Y, Makuuchi H. Focus on the conditions of resection and reconstruction in gastric cancer. What extent of resection and what kind of reconstruction provide the best outcomes for gastric cancer patients? Digestion. 2005;71(4):213-24. doi: 10.1159/000087046. Epub 2004 Sep 6. PMID 16024924